CLINICAL TRIAL: NCT02207686
Title: Assessment of Residual VHL Function in Tumors - Can it Predict the Patients' Individual Course of Disease?
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Marie Luise Bisgaard, MD (Other)
Responsible Party: Sponsor-Investigator, Marie Luise Bisgaard, MD, Associate professor, University of Copenhagen
Organization: University of Copenhagen (Other)
Other Study IDs: H-2-2010-012-A
Record Dates: First submitted 2014-08-01; First posted 2014-08-04 (Estimated); Last update posted 2015-11-13 (Estimated); Status verified 2015-11

CONDITIONS: Von Hippel-Lindaus Disease
Keywords: CNS hemangioblastoma; Renal Cell Carcinoma; VHL germline mutation; VHL somatic mutation; Tumor development
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Whole blood Tumor tissue (Paraffin embedded and fresh frozen)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- von Hippel-Lindau disease: Patients with von Hippel-Lindau disease who have had at least one vHL-related tumor removed

SUMMARY:
The investigators aim to analyze tumors from vHL patients who have different courses of disease and different types of VHL gene alterations to characterize which types of genetic alterations the tumors contain and how these alterations affect the tumor cells' behavior on a molecular level. The investigators will then compare these observations to vHL disease outcome in patients and families.

It is already known that most vHL tumors develop when both copies of the VHL gene in a cell are inactivated. The first copy is inactivated in all the person's cells from birth ("first hit"), leaving just one functional copy. A tumor can develop from cells where the second copy is also inactivated ("second hit"). So far, only the molecular consequences of the first hit have been investigated. It is our hypothesis that both the first and second hits in combination have consequences for tumor development and clinical outcome. The investigators will include tumors from patients with different disease courses and different types of "first hits" and analyse the tumors' DNA in order to find correlations between the first and second hits and patients' and families' medical histories. The investigators hereby hope to give new insights into how vHL tumors grow and which genetic factors influence tumor development. These results will contribute to the current knowledge of vHL and help us get one step closer to be able to predict an individual's tumor risks and need for surveillance.

DETAILED DESCRIPTION:
In vHL tumors from patients with different phenotypes and different genetic backgrounds, the investigators aim to assess both the nature of germline and somatic VHL mutations along with the total residual VHL protein (pVHL) activity in tumor cells and evaluate association to disease outcome in patients and families.

vHL tumor development follows Knudson's "two-hit-mode": patients are born with a germline mutation in one copy of their VHL gene in all the cells of the body - "the first hit". Somatic mutation in the other copy of the VHL gene - "the second hit" - initiates tumor development. Pheno-genotype correlations are well known in vHL, but have so far been explained exclusively by the nature of the germline mutation (the first hit). It is the investigators' hypothesis that it is the total residual activity of the protein (pVHL) present in the tumor after both first and second hit, which decides each tumor's destiny.

The investigators will apply Sanger sequencing, MLPA (and multiplex ligation dependent probe amplification), LOH (Loss of heterogeneity) analysis, methylation assays, FISH (Fluorescence In Situ Hybridization), and immunohistochemistry to characterize the germline and somatic mutations, determine presence of mRNA and pVHL, and assess residual VHL activity in each tumor. All these methods are already established in our laboratory.

The results will give deeper insight to vHL tumorigenesis and pave the road to future individual prediction of each patient´s course of disease and need for surveillance.

ELIGIBILITY:
Inclusion Criteria:

* vHL diagnosed in patient
* Patient over 18 years of age
* Informed consent to participate can be obtained
* Patient has had at least one vHL-related tumor removed
* A reference DNA sample (from blood or normal tissue) and tumor tissue (paraffin-embedded or fresh frozen) can be obtained.

Exclusion Criteria:

* Patients under the age of 18 years
* Patients who had not previously had a vHL-related tumor removed
* Patients whos previously removed tumor tissue cannot be obtained or is of such a quantity or quality that no exact histological analysis can be done and/or no DNA can be extracted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: vHL patients over 18 years of age who have had at least one vHL-related tumor removed, and for whom a reference DNA sample (from blood or normal tissue) and tumor tissue (paraffin-embedded or fresh frozen) can be obtained.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Residual pVHL activity measured by amount of VHL mRNA in tumor cells | Two years
  We will correlate amount of VHL mRNA in tumor cells with the type of the patients' first hit (germline mutation) and the tumor's second hits (somatic mutations).

SECONDARY OUTCOMES:
Presence of VHL protein (pVHL) in tumor cells | Two years
  We will correlated the presence of pVHL in tumor cells with the nature of the patients' (germline mutation) and the tumor cells' second hits (somatic mutations).
Type of second hit (somatic mutation) found in DNA from tumor cells | One year
  We will correlate the type of germline mutation found in the patient's DNA from blood with the types of second hits (somatic mutations) found in the tumor's DNA.
Patient's age at tumor diagnosis | Two years
  For each tumor we will correlate the previous outcome measures to the patient's age at tumor diagnosis
Patient's total tumor burden | Two years
  For each tumor we will correlate the previous outcome measures to the patient's total tumor burden

OTHER OUTCOMES:
Type of clinical vHL in the patient's family (e.g. type 1, type 2) | Two years
  For each tumor we will correlate the previous outcome measures to the type of clinical vHL found in the patient's family.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Luise Bisgaard, MD, Principal Investigator — Department of Cellular and Molecular Medicine, University of Copenhagen
Locations (1):
- Department of Cellular and Molecular Medicine, University of Copenhagen, Copenhagen, Copenhagen N, Denmark